CLINICAL TRIAL: NCT00425074
Title: Pharmacodynamic- Pharmacokinetic Trial, Comparative Double Blind, of the Chronic Administration of 150 mg of Slow Release ASA Versus 150 mg of Normal Release ASA, in the Platelet Functionalism.
Brief Title: Pharmacodynamic-pharmacokinetic Trial, of Slow Release ASA, in the Platelet Functionalism.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rottapharm Spain (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TROM-EC-ECC-FIb
Record Dates: First submitted 2007-01-19; First posted 2007-01-22 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Cardiovascular Disease
Keywords: slow release ASA; platelet functionalism; secondary cardiovascular prevention
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- SR-ASA (Experimental): slow release acetylsalicylic acid 150 mg
  Interventions: Drug: slow release acetyl salicylic acid; Drug: SR-ASA
- ASA (Active Comparator): normal release acetylsalicylic acid
  Interventions: Drug: ASA

INTERVENTIONS:
Drug: slow release acetyl salicylic acid — 150 mg in capsules via oral, during 14 days.
  Arms: SR-ASA
Drug: ASA — normal release acetylsalicylic acid
  Arms: ASA
Drug: SR-ASA — slow release acetylsalicylic acid 150 mg
  Arms: SR-ASA

SUMMARY:
The purpose of this study is to evaluate the platelet antiaggregant effect that a chronic treatment with ASA (150 mg) produces,comparing this effect between two formulations of ASA: normal and the one of sustained release, in patients with stable coronary disease.

DETAILED DESCRIPTION:
A large clinical trials have established the efficacy of the antiaggregant products in patients with ischemic cardiopathy, stroke and intermittent claudication.

Without doubt, the acetylsalicylic acid (ASA) is the most used antiaggregant product, nevertheless, and spite of being centenarian, it last some questions pending regarding the most appropriate dose, mechanism of action implicated, the association with other drugs, and the pharmaceutical form in order to improve the efficacy and the safety of the ASA.

Some previous studies indicate that the slow release form of ASA has a different behaviour in the platelet effect in comparison with plain formulation.

The aim of this study is to demonstrate the best antiaggregant and safety profile of a low dose of a slow release formulation of ASA.

ELIGIBILITY:
Inclusion Criteria:

* Previous episodes of myocardial infarction
* Previous episodes of instable angina pectoris
* Previous coronary revascularization
* Significant arterial coronary disease

Exclusion Criteria:

* Patients with other pathologies that requires treatment with other antiaggregants
* Patients in treatment with low molecular weight heparin or oral anticoagulant
* Patients with antecedents of hypersensibility to ASA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-01; Primary Completion 2007-06 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of the treatment with ASA (150 mg) produces on the thromboxan/prostacyclin balance and its repercussion in the platelet aggregation,comparing this effect between two formulations | 28 days

SECONDARY OUTCOMES:
To evaluate the principal kinetic parameters of both galenic formulations of ASA. | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Eloy Rueda, MD, Principal Investigator — Hosp. Universitario Virgen de la Victoria, Málaga (Spain); José Pedro de la Cruz, PhD, Principal Investigator — Departmento de Farmacología y Terapéutica Clínica Facultad de Medicina, Universidad de Málaga; José Antonio González Correa, PhD, Principal Investigator — Departamento de Farmacología y Terapéutica Clínica Facultad de Medicna, Universidad de Málaga
Locations (1):
- Hospital Universitario Virgen de la Victoria, Málaga, Spain